CLINICAL TRIAL: NCT06100887
Title: A Phase 2 Study to Evaluate the Effect of EDG-5506 on Safety, Pharmacokinetics, and Biomarkers in Children and Adolescents With Duchenne Muscular Dystrophy Previously Treated With Gene Therapy
Brief Title: Phase 2 Study of EDG-5506 in Children and Adolescents With Duchenne Muscular Dystrophy Previously Treated With Gene Therapy
Acronym: FOX
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Edgewise Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDG-5506-215
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 1; Drug: Placebo
- Cohort 2 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 2; Drug: Placebo
- Cohort 3 (Experimental): Drug: Sevasemten Drug: Placebo
  Interventions: Drug: Sevasemten Dose 3; Drug: Placebo

INTERVENTIONS:
Drug: Sevasemten Dose 1 — Sevasemten is administered orally once per day
  Arms: Cohort 1
Drug: Sevasemten Dose 2 — Sevasemten is administered orally once per day
  Arms: Cohort 2
Drug: Sevasemten Dose 3 — Sevasemten is administered orally once per day
  Arms: Cohort 3
Drug: Placebo — Placebo is administered orally once per day

SUMMARY:
The FOX study is a 2-part, multicenter, Phase 2 study of safety, pharmacokinetics, and biomarkers in children and adolescents with Duchenne muscular dystrophy previously treated with gene therapy including a randomized, double-blind, placebo-controlled Part A, followed by an open-label part B.

DETAILED DESCRIPTION:
FOX is a 2-part, multi-center, Phase 2 study to evaluate the effect of sevasemten (EDG-5506) on safety, pharmacokinetics and biomarkers of muscle damage in approximately 48 children and adolescents with Duchenne muscular dystrophy treated with oral, once-daily sevasemten. This study will have up to a 4-week Screening period, a 12-week randomized double-blind, placebo-controlled treatment period (Part A), followed by up to a 144-week open-label extension period (Part B).

Approximately forty-eight (48) participants aged 6 to 17, inclusive, will be randomized to sevasemten or placebo in a 2:1 ratio. Three dose cohorts (Cohort 1, Cohort 2 and Cohort 3) of approximately 12 participants each will be enrolled. Approximately 12 additional participants may be added to 1 of these cohorts.

After review of emerging data, the protocol was amended so all dose cohorts receive the same dose in Part B.

ELIGIBILITY:
Key Inclusion Criteria:

* Aged 6 to 17 with a documented mutation on the DMD gene and phenotype consistent with DMD.
* Prior receipt of an AAV-based gene therapy (≥ 2 years after documented receipt of gene therapy administration or ≥ 3 years after randomization in a randomized study).
* Able to complete stand from supine in ≤ 8 seconds at the Screening visit and able to perform the 4-stair climb in < 10 seconds at the Screening visit.
* Body weight ≥ 15 kg at the Screening visit.
* Treatment with a stable dose of corticosteroids for a minimum of 6 months prior to the Baseline visit.

Key Exclusion Criteria:

* Medical history or clinically significant physical exam/laboratory result that, in the opinion of the investigator, would render the participant unsuitable for the study. This includes venous access that would be too difficult to facilitate repeated blood sampling.
* Screening visit cardiac echocardiography showing left ventricular ejection fraction (LVEF) < 40%.
* Receipt of an investigational drug (other than the AAV-based gene therapy per Inclusion criteria) within 30 days or 5 half-lives (whichever is longer) of the Screening visit in the present study.
* Receipt of an exon-skipping therapy within 6 months prior to the Screening visit.

Ages: 6 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events during treatment with sevasemten or placebo | 36 months
  All participants
Severity of adverse events during treatment with sevasemten or placebo | 36 months
  All participants

SECONDARY OUTCOMES:
Incidence of laboratory test-related treatment emergent adverse events | 36 months
  All participants
Pharmacokinetics as measured by steady state plasma concentration | 36 months
  All participants
Change from Baseline in serum creatine kinase | 12 weeks
  All participants
Change from Baseline in fast skeletal muscle troponin I | 12 weeks
  All participants

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - UCLA Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Florida, Gainesville, Florida
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rare Disease Research, Hillsborough, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor Website — http://edgewisetx.com